CLINICAL TRIAL: NCT04208542
Title: Effects of Thoracic Erector Spinae Plane Blockade on Acute and Chronic Pain After Video Assisted Thoracoscopic Surgery (VATS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2019-0050
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Thoracic
Keywords: Thoracic surgical procedures

STUDY DESIGN:
Intervention Model Description: 2 groups of patients will be studied simultaneously. One group will have the intervention of the ESP block and IV PCA. The other group will have only IV PCA.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both participants and anesthesia provider will not know which intervention applied. Another anesthesia provider who did not perform nerve block will follow and record to the study data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Active Comparator): Under general anaesthesia, ultrasound guided ESP block will perform at the T5 level with 0.375% ropivacaine 20ml. Fentanyl 1 ug/kg will administer at last 30 minutes of surgery for postoperative analgesia. Patient controlled analgesia (PCA) with fentanyl (10 ug/kg) and palonosetron 0.075mg will apply to the all patients. Postoperative pain assessment and opioid consumption will record till the postoperative 48 hours. Pain assessment will record 3 months after surgery.
  Interventions: Drug: ESP block
- Control (No Intervention): Fentanyl 1 ug/kg will administer at last 30 minutes of surgery for postoperative analgesia. Patient controlled analgesia (PCA) with fentanyl (10 ug/kg) and palonosetron 0.075mg will apply to the all patients. Postoperative pain assessment and opioid consumption will record till the postoperative 48 hours. Pain assessment will record 3 months after surgery.

INTERVENTIONS:
Drug: ESP block — Ultrasound guided Erector spinae block (ESP) will perform.
  Arms: Interventional

SUMMARY:
This is a prospective randomized study intended to assess the efficacy of erector spinae plane analgesia on acute and chronic postoperative pain for VATS procedures. It will include 72 patients presenting to Severance hospital for a VATS procedure. Patients will be randomized 1:1 to receive either ESP block and intravenous patient-controlled analgesia (IV PCA) or IV PCA only. Ropivacaine will be used in nerve block, and injected at the end of surgery. The primary outcome will be to compare analgesic efficacy between the two groups as defined by immediate postoperative pain scores on the numeric pain rating scale. Secondary outcomes include total opioid consumption, painDETECT score, and chronic pain scores.

DETAILED DESCRIPTION:
Postoperative pain control for thoracic surgery is key to allow faster recovery and diminish postoperative complications. Poorly controlled acute pain may contribute to the impairment of respiratory function and the development of chronic post-thoracotomy pain.

Recently, an increasing number of erector spinae plane (ESP) nerve blocks are being performed as it has been demonstrated, and via case reports that the blocks provide clinical effectiveness, but may have a better side-effect profile than the paravertebral nerve block and epidural analgesia. Moreover, there is an advantage for novice because ESP block is simpler and safer to proceed than conventional nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female participants providing written informed consent,
2. ASA grade 1-3,
3. aged over 20 and under 80,
4. primary lung cancer participants scheduled segmentectomy or lobectomy c MLND,
5. undergoing a VATS procedure under General Anaesthesia

Exclusion Criteria:

1. Absence of informed written consent,
2. chemotherapy before or after surgery,
3. pre existing infection at block site,
4. severe coagulopathy,
5. pre existing neurological deficit,
6. previous history of opiate abuse,
7. pregnancy,
8. pre existing chronic pain condition,

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | up to postoperative 48 hours.
  These scores will record till the postoperative 48 hours.
  - The Numerical Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
opioid consumption | postoperative 48th hours
  Total opioid consumption will calculate and record till the postoperative 48th hours.
opioid consumption | 3 months after surgery.
  Total opioid consumption will calculate and record till the postoperative 3 months after surgery.
postoperative painDETECT score | up to postoperative 3 months.
  painDETECT is a nine-item questionnaire that consists of seven sensory symptom items for pain that are graded from 0= never to 5= strongly, one temporal item on pain-course pattern graded -1 to +1, and one spatial item on pain radiation graded 0 for no radiation or +2 for radiating pain.
NRS | up to postoperative 3 months.
  NRS will record at postoperative 3 months.
  - The Numerical Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea